CLINICAL TRIAL: NCT06467604
Title: CRAVE Study: Comparing Craving Responses and Diet Quality of GLP1 Receptor Agonist Users
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Knownwell (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2184712
Record Dates: First submitted 2024-06-11; First posted 2024-06-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: GLP-1; diet quality; weight loss; anti-obesity medication; food cravings
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Surveys and Questionnaires; Diet Records; Calorimetry, Indirect; Body Composition; Waist Circumference; Body Height; Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Semaglutide: eligible patients who are prescribed semaglutide for their obesity-management
  Interventions: Behavioral: Surveys; Other: Indirect Calorimetry; Other: Body composition; Other: Anthropometrics
- Tirzepatide: eligible patients who are prescribed tirzepatide for their obesity-management
  Interventions: Behavioral: Surveys; Other: Indirect Calorimetry; Other: Body composition; Other: Anthropometrics

INTERVENTIONS:
Behavioral: Surveys — Participants will be provided electronic surveys at 3 timepoints throughout study.
  Other Names: FCI-II; 3 day Food Diary; Hunger VAS; BED-7; HFSS 2-item food insecurity survey; MESA Neighborhood Healthy Food
Other: Indirect Calorimetry — Participants will receive indirect calorimetry at 3 time points throughout the study.
Other: Body composition — Participants will receive body scans using bioelectrical impedence seca mBCA 554 digital body composition analysis scale 3 time points throughout the study.
  Other Names: Seca mBCA 554
Other: Anthropometrics — Participants will have their Height, weight, waist circumference, and calculated BMI performed at 3 time points throughout the study.
  Other Names: Waist circumference; Height; Weight

SUMMARY:
This study aims to assess the impact of GLP-1 receptor agonists, semaglutide and tirzepatide, on food cravings and diet quality in individuals with overweight or obesity. Over 24 weeks, up to 150 adult participants will be monitored using questionnaires and dietary records at 0, 12, and 24 weeks to measure changes in diet quality, disordered eating, food cravings, and hunger. This research, conducted with Seen Medical Group at Knownwell Health Clinic, seeks to fill the gap in literature on the dietary quality effects of GLP-1RAs.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of GLP-1 receptor agonist (GLP-1RA) medications, specifically semaglutide and tirzepatide, on food cravings and diet quality among individuals diagnosed with overweight and obesity. Participants will be recruited through Knownwell Health clinical staff, who will refer eligible patients to the UCD research team for further information and screening.

At Knownwell Clinic, standard care for patients on GLP-1RA medications includes blood draws, blood pressure evaluations, body composition analysis (Seca), and indirect calorimetry testing. These procedures will be conducted at baseline (week 0), midpoint (weeks 8-12), and end of titration/max dose (week 24).

Participants will complete a series of virtual questionnaires on nutrition, eating habits, and diet quality, along with a 3-day food diary. Regular medical appointments will follow Knownwell Clinic's standards of care. Participants must procure their own GLP-1RA medication. This study adds questionnaires to assess: dietary quality (photo-based food records), hunger (hunger VAS survey) and food cravings (FCI-II) related to GLP-1RA use.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18.0-<70 years
2. Obese (BMI greater than or equal to 30.0 kg/m2) or overweight (BMI greater than or equal to 27.0 kg/m2) with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension, dyslipidemia, obstructive sleep apnea or cardiovascular disease and history of at least one self-reported unsuccessful dietary effort to lose body weight will be recruited.
3. On stable regimen of medications that can affect weight or diabetes outcomes for at least 3 months (brief regimens of medications such as antibiotics, steroids, etc. are permitted)
4. Weight stable (+/- 5%) over previous 3 months
5. Be under the care of a physician who will be responsible for managing participant's treatment regimen
6. Willingness to provide food diary data throughout trial
7. Access to a smartphone/tablet that can download the food logging application
8. Willing and able to provide a valid email address for use in the study
9. Be able to communicate (oral and written) in English
10. Be able to provide informed consent

Exclusion Criteria:

1. History of weight loss surgery
2. History of major surgery within three months of enrollment
3. Recent weight fluctuations exceeding 5 kg within a 3-month period preceding screening
4. Use of systemic hormonal therapies (contraceptive medication is allowed)
5. History of Type 1 or type 2 diabetes, HgbA1c ≥ 6.5% (gestational diabetes is allowed)
6. Hemoglobinopathy that interferes with measurement of HbA1c
7. Treatment with any GLP-1 Receptor Agonist medication(s) within 90 days of screening
8. Significant kidney or liver disease, malnutrition, or any condition that, in the investigator's judgment, should exclude participation
9. Documented chronic diseases including thyroid disease, kidney disease, active cancer, previous cardiovascular events, history or presence of chronic pancreatitis, or other gastrointestinal issues
10. Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
11. Current cancer or cancer treatment, or history of cancer or cancer treatment within the last 3 years, excluding specific cases
12. Diagnosis or strong clinical suspicion of eating disorders
13. Background of significant active or unstable major depressive disorder (MDD) or any other severe psychiatric disorder within the past 2 years
14. Lifetime history of a suicide attempt
15. History of gastroparesis or other gut dysmotility syndrome
16. Prior use of other GLP-1RA or combination GIP/GLP-1RA medications or previous participation in any GLP-1RA trials
17. Pregnant or lactating women, women planning to become pregnant in the next 12 months
18. Multiple patient-reported food allergies/intolerances significantly limiting food intake
19. Smoking, illicit drug use, vaporizer and/or electronic cigarette use
20. Currently consuming >14 alcoholic drinks per week
21. Extreme dietary or exercise patterns
22. Individuals who are not yet adults (infants, children, teenagers)
23. Individuals who are currently incarcerated or serving a prison sentence
24. Individuals unable to provide informed consent due to factors such as mental incapacity or language barriers
25. Any disorder, inability, or unwillingness to comply with the study protocol that may jeopardize patient safety or compliance, based on the investigator's opinion

Pregnancy and Other Exclusions during Trial:

1. If a patient experiences a pregnancy, her data will be censored from the time of estimated conception, and she will be excluded from further participation.
2. If a patient develops active cancer (except skin cancer), they will be excluded from further participation due to safety concerns/contraindications for weight loss.
3. If a patient develops another exclusionary condition, such as unstable angina or another condition for which weight loss or exercise might be contraindicated, further participation will be determined by the Medical Monitoring Team (PI, Project Manager).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes male and female participants aged 18 to under 70 years diagnosed with obesity (BMI ≥ 30 kg/m²) or overweight (BMI ≥ 27 kg/m²) with at least one weight-related comorbidity (e.g., hypertension, dyslipidemia, sleep apnea, cardiovascular disease). They must have a history of at least one unsuccessful dietary effort to lose weight and be on a stable medication regimen affecting weight or diabetes outcomes for at least three months. Short courses of antibiotics and steroids are allowed. Participants must have maintained a stable weight (±5%) over the past three months, be under physician care, provide food diary data, have a smartphone or tablet for a food logging app, communicate in English, and provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Food Craving Score | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
  Effect of GLP1 medications on food cravings measured by the food-craving inventory (FCI-II) questionnaire.The FCI-II is scored on a Likert scale from 1-5, with 1 being "Never," 5 being "Always/Almost every day."

SECONDARY OUTCOMES:
Change in USDA Healthy Eating Index-2015 (HEI) Score | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
  Effect of GLP1 medications on Healthy Eating Index-2015. The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations and dietary patterns published in the Dietary Guidelines.

OTHER OUTCOMES:
Changes in weight in kilograms | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
  Effect of GLP1 medications on weight (in kg)
Changes in waist circumference (cm) | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
Changes in resting metabolic rate (RMR) | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
  Effect of GLP1 medications on resting metabolic rate, assessed by indirect calorimetry.
Change in weight loss percentage | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
Changes in body fat percentage | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
  Measured by seca mBCA 554 bioelectrical impedance analysis
Changes in skeletal muscle mass (lbs) | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
  Measured by seca mBCA 554 bioelectrical impedance analysis
Changes in visceral fat mass (L) | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
  Measured by seca mBCA 554 bioelectrical impedance analysis
Changes in segmental skeletal muscle mass (lbs) | Baseline, Midpoint (8-12 weeks), End of study (24 + 2 weeks)
  Measured by seca mBCA 554 bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Knownwell, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No